CLINICAL TRIAL: NCT02188264
Title: A Phase IB Study of the Combination of AZD6244 Hydrogen Sulfate (Selumetinib) and Cyclosporin A (CsA) in Patients With Advanced Solid Tumors With an Expansion Cohort in Metastatic Colorectal Cancer
Brief Title: Selumetinib and Cyclosporine in Treating Patients With Advanced Solid Tumors or Advanced or Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-01484; NCI-2014-01484 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 13-2628; 9571 (Other: University of Texas MD Anderson Cancer Center LAO); 9571 (Other: CTEP); K23CA190849 (NIH); P30CA016672 (NIH); UM1CA186644 (NIH); UM1CA186686 (NIH); UM1CA186688 (NIH); UM1CA186690 (NIH); UM1CA186704 (NIH); UM1CA186709 (NIH); UM1CA186712 (NIH); UM1CA186716 (NIH); UM1CA186717 (NIH)
Record Dates: First submitted 2014-07-10; First posted 2014-07-11 (Estimated); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Recurrent Colorectal Carcinoma; Solid Neoplasm; Stage IIIA Colorectal Cancer AJCC v7; Stage IIIB Colorectal Cancer AJCC v7; Stage IIIC Colorectal Cancer AJCC v7; Stage IVA Colorectal Cancer AJCC v7; Stage IVB Colorectal Cancer AJCC v7
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cyclosporine; Cyclosporins; AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (selumetinib and cyclosporine) (Experimental): Patients receive selumetinib PO BID on day -7 of course 1 and then on days 1-28 (one dose on day 1 only). Patients also receive cyclosporine PO BID on day -3 of course 1 and then on days 1-28 (one dose on day 1 only). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclosporine; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Selumetinib

INTERVENTIONS:
Drug: Cyclosporine — Given PO
  Other Names: 27-400; Ciclosporin; CsA; CyA; Cyclosporin; Cyclosporin A; Cyclosporine Modified; Gengraf; Neoral; OL 27-400; Sandimmune; SangCya
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Selumetinib — Given PO
  Other Names: ARRY-142886; AZD 6244; AZD-6244; AZD6244; MEK Inhibitor AZD6244

SUMMARY:
This phase I/Ib trial studies the side effects and best dose of selumetinib when given together with cyclosporine in treating patients with solid tumors or colorectal cancer that have spread to other places in the body and cannot be cured or controlled with treatment. Selumetinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Biological therapies, such as cyclosporine, use substances made from living organisms that may stimulate or suppress the immune system in different ways and stop tumor cells from growing. Giving selumetinib and cyclosporine may be a better treatment for solid tumors or colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of the combination of AZD6244 (selumetinib) and cyclosporin A (cyclosporine) in adult patients with advanced solid tumors.

SECONDARY OBJECTIVES:

I. To determine the safety profile and tolerability of this regimen in this patient population.

II. To determine the pharmacokinetics of the combination. III. To evaluate the selected biomarkers of drug effect in patients with advanced solid tumors or refractory metastatic colorectal cancer (CRC).

IV. Evaluate the activity of the combination in terms of objective response rate (per Response Evaluation Criteria in Solid Tumors [RECIST] 1.1), progression-free survival (PFS).

OUTLINE: This is a phase I, dose-escalation study of selumetinib followed by a phase Ib study.

Patients receive selumetinib orally (PO) twice daily (BID) on day -7 of course 1 and then on days 1-28 (one dose on day 1 only). Patients also receive cyclosporine PO BID on day -3 of course 1 and then on days 1-28 (one dose on day 1 only). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Before any study procedures are performed, subjects will have the details of the study described to them, and they will be given a written informed consent document to read; then, if subjects consent to participate in the study, they will indicate that consent by signing and dating the informed consent document in the presence of study personnel
* DOSE ESCALATION PHASE: Histological or cytopathological diagnosis of an advanced cancer that is refractory to standard therapy or for which no standard therapy exists
* COHORT EXPANSION PHASE: Histological or cytopathological diagnosis of advanced/metastatic unresectable colorectal cancer with known rat sarcoma viral oncogene homolog (RAS) mutational status; patients with known B-Raf proto-oncogene, serine/threonine kinase (BRAF) mutations will not be eligible for the expansion cohort; all patients must have received and progressed or be intolerant of an oxaliplatin-containing regimen and an irinotecan-containing regimen
* COHORT EXPANSION PHASE: At least one tumor lesion amenable to core needle biopsy without unacceptable risk of a major procedural complication (one pretreatment and at least one on-treatment biopsy will be performed)
* COHORT EXPANSION PHASE: Patient must have measurable lesions as defined by RECIST version 1.1 criteria
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Estimated life expectancy > 3 months
* Absolute neutrophil count (ANC) >= 1,500/mcl
* Platelets >= 100,000/mcl
* Hemoglobin >= 9 g/dl
* Estimated glomerular filtration rate (eGFR) greater than or equal to 60 ml/min/1.73 m^2
* Serum total bilirubin < 1.5 x upper limit or normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]), alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN; if liver involvement, AST, ALT =< 5.0 x ULN
* Alkaline phosphatase =< 2.5 x ULN; if liver involvement, alkaline phosphatase =< 5.0 x ULN
* Serum albumin >= 2.5 g/dl
* International normalized ratio (INR) =< 1.5 x ULN or prothrombin time (PT) =< 1.5 x ULN seconds above control unless patient is currently receiving warfarin therapy for the treatment or prevention of venous thrombosis
* A male subject of fathering potential must use an adequate method of contraception to avoid conception throughout the study (and for up to 12 weeks after the last dose of study drug) to minimize the risk of pregnancy; if the partner is pregnant or breastfeeding, the subject must use a condom
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 12 weeks after the last dose of study drug to minimize the risk of pregnancy; WOCBP must have a negative serum or urine pregnancy test within 72 hours before the start of the investigational product
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients who are receiving any other investigational agents
* Prior full field radiotherapy < 4 weeks or limited field radiotherapy < 2 weeks prior to first study drug administration
* Patients with brain metastases may participate in this trial provided they are clinically stable; patients who are < 1 month from definitive therapy, receiving steroid therapy or taper, or anti-convulsant medications (started for brain metastases) must not be included
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to AZD6244 or cyclosporine A or their excipients
* Patients with a history of thrombotic or embolic events within the last six months such as a cerebrovascular accident (including transient ischemic attacks), pulmonary embolism
* Cardiac conditions as follows:

  * Active coronary artery disease, unstable or newly diagnosed angina or myocardial infarction less than 12 months prior to first study drug administration
  * Class II-IV New York Heart Association (NYHA) congestive heart failure
  * Uncontrolled hypertension (systolic blood pressure [BP] > 150 mmHg and diastolic BP > 90 mmHg for 24 hours) despite optimal medical management; blood pressure must be below 140/90 mmHg at screening; subjects with a history of hypertension who are receiving treatment with calcium channel blockers that are cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) substrates should be changed to an alternative antihypertensive medication prior to first study drug administration
  * Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin
  * Corrected QT (QTc) (Frederica) prolongation > 480 msec
  * Subjects with valvular heart disease Common Terminology Criteria for Adverse Events (CTCAE) (version 4.0) grade 2
  * Known left ventricular ejection fraction (LVEF) < 50%
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris (Canadian Cardiovascular Society grade II-IV despite medical therapy), cardiac arrhythmia, active bleeding diatheses, or psychiatric illness/social situations that would limit compliance with study requirements
* Known ophthalmological conditions as follows: intra-ocular pressure > 21 mmHg, or uncontrolled glaucoma (irrespective of intra-ocular pressure); current or past history of central serous retinopathy or retinal vein occlusion
* Major surgical procedure, open biopsy, or significant traumatic injury less than 3 weeks or those who receive minor surgical procedures (eg core biopsy or fine needle aspiration) within 1 week from first dose of first study drug administration
* Known inability to swallow capsules
* Known history of human immunodeficiency virus (HIV), hepatitis B, and/or hepatitis C (no additional laboratory tests for HIV, hepatitis [Hep] B, or Hep C are required for screening)
* Inability to comply with study and/or follow-up procedures
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with AZD6244
* Patients with hyponatremia (sodium < 130 mmol/L)
* Baseline serum potassium < 3.5 mmol/L (potassium supplementation may be given to restore the serum potassium above this level prior to study entry)
* Baseline serum calcium < 8.4 mg/dL (calcium supplementation may be given to restore the serum calcium above this level prior to study entry)
* Prisoners or subjects who are involuntarily incarcerated
* Patients who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-08-29 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
Incidence of DLT defined as any grade 3 non-hematological toxicity or grade 4 hematological toxicity attributed to selumetinib or cyclosporine graded per National Cancer Institute (NCI) CTCAE version 4.0 | 28 days
  The maximum tolerated dose will be defined as the highest dose in which 0 or 1 out of 6 patients have a DLT.

SECONDARY OUTCOMES:
Incidence of adverse events that occur after course 1, day 1 assessed using NCI CTCAE version 4.0 | Up to 30 days after completion of study treatment
  Adverse events will be tabulated by type and grade.
Pharmacokinetic (PK) parameters, including the distribution of area under the curve and maximum concentration | Pre-dose, 0.5, 1, 2, 4, 8, and 24 hours on days -7, -3, and 1 of course 1
  Looking at historical data on patients previously treated on single-agent therapy, the distribution of these PK parameters will be estimated in patients treated with single-agent selumetinib and single-agent cyclosporine. The distribution of these parameters in the combination study will be qualitatively compared to the single-agent distribution.
Objective tumor response based on computed tomography scans (or magnetic resonance imaging if patients are allergic to iodinated contrast) per RECIST 1.1 criteria | Up to 30 days after completion of study treatment
  Analysis of efficacy measures will be descriptive. Antitumor activity of the combination of selumetinib and cyclosporine will be based on the best overall response. Response rate (complete response [CR], partial response [PR], CR + PR) will be tabulated with 95% exact binomial confidence intervals. If applicable, response rate will also be tabulated by patients' baseline gene mutation status (eg, KRAS and BRAF). Data listings will present disease response category (eg, CR, PR, stable disease), duration of response, and as appropriate, tumor marker measurements.
Progression-free survival (PFS) | From first therapy received to documented disease progression or death from any cause, assessed up to 30 days after completion of study treatment
  PFS will be estimated using the product-limit method of Kaplan and Meier.

OTHER OUTCOMES:
Change in expression of phosphorylated-mitogen-activated protein kinase 1 | Baseline to up to 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Christopher H Lieu, Principal Investigator — University of Texas MD Anderson Cancer Center LAO
Locations (10):
- United States (9):
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada